CLINICAL TRIAL: NCT04859309
Title: Activating Older People After a Hip Fracture
Acronym: ActiveHip
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Amgen (Industry); Institut de formació contínua - IL3 (Unknown); University of Barcelona (Other); Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other); EIT Health (Other); Biohealth Research Institute in Granada (ibs.GRANADA) (Unknown)
Responsible Party: Principal Investigator, Patrocinio Ariza Vega, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Andalusian Health System
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Hip Fractures
Keywords: Tele-rehabilitation; Occupational therapy; Physiotherapy; Physical exercise; Function; Quality of life; Informal Caregiver burden; Information and Communication Technologies
MeSH Terms: conditions — Hip Fractures; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ActiveHip Intervention (Experimental): The ActiveHip tele-rehabilitation mobile application.
  The program consists of a multidisciplinary home-based tele-rehabilitation program delivered through a mobile application. It is comprised by an occupational therapy program and a physical exercise program.
  The intervention group have the opportunity to perform three online-based sessions per week (two sessions of physical exercise and one of occupational therapy), each lasting 30-60 min. It is able to realize a fourth session, called "bonus session".
  In addition, the intervention group will receive the educational program, which has a total of 7 modules. 5 modules are for patients and caregivers, and 2 modules are specific for caregivers.
  Interventions: Behavioral: ActiveHip+ mobile application
- Standard care (Active Comparator): Participants of this group will receive the standard care for hip fracture patients at hospital discharge.
  Interventions: Procedure: Standard care in a hip fracture

INTERVENTIONS:
Behavioral: ActiveHip+ mobile application — The mobile application with the educational and multidisciplinary tele-rehabilitation program.
  Arms: ActiveHip Intervention
Procedure: Standard care in a hip fracture — The participants of this group will receive the standard treatment for a hip fracture in the Andalusian healthcare system.
  Arms: Standard care

SUMMARY:
The main aim of this study is to determine if the ActiveHip tele-rehabilitation mobile application improves the functional level and the quality of life of patients who undergone hip surgery after a fracture.

The second aim is to determine if the ActiveHip intervention reduce the anxiety, stress and burden of the caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Have hip fracture surgery
* Age equal to or greater than 65 years
* Are allowed weight-bearing at 48 hours after surgery
* Had a high pre-fracture functional level the week before the fracture (Functional Independence Measure [FIM] index scored more than 90 points)
* Have an informal or family caregiver who has the ability to access the Internet to use the app ActiveHip+
* Basic management of the mobile phone
* Have signed an informed consent.

Exclusion Criteria:

* Presence of low cognitive level (Pfeiffer test score lower than 4 points)
* Being dependent on the activities of daily living before the hip (Functional Independence Measure [FIM] index scored less than 60 points)
* Being institutionalized
* Post-surgery complications
* Terminal disease
* Age under 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | The primary outcome will be followed over 12 weeks.
  The SPPB is one of the most commonly used instruments for measuring physical performance in population studies. The SPPB assessment has previously been used to evaluate the mobility of older people and patients with a hip fracture. The performance battery consists of three tasks: balance, walking, and chair stands. The SPPB tests of balance, including time to walk 4 meters and time required to stand from a chair 5 times. The score ranges from 0 to 12 points, with higher scores indicating better mobility. Low scores on the SPPB have a high predictive value for a wide range of health consequences including disability in Activities of Daily Living, loss of mobility, disability, hospitalization duration of stay in the hospital, admission to nursing facilities, and death. Internal consistency is high, with Cronbach's α = 0.87.

SECONDARY OUTCOMES:
EuroQoL 5D Quality of Life questionnaire | 12 weeks
  The EuroQol (EQ-5D) is a patient-reported outcome measure used to evaluate the generic quality of life of the patient. The questionnaire comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 possible levels: no problems, some problems, and extreme problems. To obtain a total score index, the EuroQol Group provides a calculator called "EQ-5D-5L Crosswalk Index Value Calculator" which is based on several studies conducted in 6 different countries (Spain among them). Additionally, it includes the EQ visual analog scale (EQ-VAS) in which the patients self-rated her/his health on a vertical analog scale from 0 (the worst health status) to 100 (the best health status).
Functional Independence Measure | 12 weeks
  The Functional Independence Measure score reflects the level of assistance a person needs in activities of daily living. The measure consists of 18 items, of which 13 concern physical activities divided into four categories: self-care, sphincter control, mobility, and locomotion. The remaining five items relate to aspects of cognitive and social functioning divided in two categories: communication and social cognition. The total functional independence measure score range is between 18 and 126 points. Higher scores indicate a higher level of independence.
Short Falls Efficacy Scale-International (SFES-I) | 12 weeks
  The SFES-I test is used to evaluate patients' fear of falling when performing ADLs. The scale consists of seven items with four possible answers corresponding to the level of concern. The total score range is from 7 to 28 points, with a higher score indicating a higher level of fear of falling. The internal consistency of the SFES-I is very high with Cronbach's α = 0.92.
New Mobility Score (NMS) | 12 weeks
  The New Mobility Score (NMS) is an easy-to-administer measure of functional ability and is used worldwide as a hip fracture (HF) score. The NMS consists of three questions to measure walking mobility across daily life activities; Indoor walking, outdoor walking; and walking during shopping which evaluates the pre-fracture functional level with a score from 0 (not able to walk) to 9 (fully independent). The inter-tester reliability of the New Mobility Score is very high and can be recommended to evaluate the pre-fracture functional level in patients with acute hip fracture. The internal consistency of the NMS is good with Cronbach's α, closer to 1.
The Short Portable Mental State Questionnaire (SPMSQ) of Pfeiffer | 12 weeks
  The SPMSQ this test has 10 items that assess various functions: orientation, recall memory, concentration, and calculation. Very brief but with an acceptable discriminatory capacity. The SPMSQ test has good reliability and validity. For clinical use, a cut-off of 3 appears to be most useful. When illiterate patients are assessed, it is recommended to employ a cut-off of 4 or more. The internal consistency of the SPMSQ is good with Cronbach's α, = 0,82.
Visual Analogue Scale for Pain (VAS Pain) | 12 weeks
  The VAS Pain test is a fast and convenient way to evaluate the intensity of pain perceived by the patient. The patient indicates the perceived pain by pointing out on a physical scale a value from 0 (without pain) to 10 (maximum pain) (Boonstra, Schiphorst Preuper, Reneman, Posthumus, & Stewart, 2008). The test-retest reliability is good with r = 0.71 for illiterate patients and r = 0.94 for literate patients.
The Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  The HADS is administered to assess the presence of anxiety and depression in both patients and caregivers. The scale consists of 14 items, each with four possible answers (0-3 points), divided into two subscales: seven items for the status of depression and the remaining items for the presence of anxiety. The maximum score of each subscale is 21 points, with scores below 11 indicating the presence of depression or anxiety. The internal consistency of the HADS is good with Cronbach's α = 0.80.
International Fitness Scale (IFIS) | 12 weeks
  The IFIS is a simple evaluation scale consisting of five questions concerning the patient's perception of his/her general physical condition (cardio-respiratory fitness, muscular strength, agility, and flexibility). Each question has five possible answers (very poor, poor, average, good, and very good) scored from 1 to 5 points, with the highest score corresponding to the best perception of physical condition. The test-retest reliability of the IFIS, as measured by the average weighted Kappa, is 0.45.
Zarit Burden Interview | 12 weeks
  The Zarit Burden Interview assessment includes 22 questions related to aspects of caregiver burden, including mood, physical state, economic situation, and social state, as well as the feelings of the caregiver when giving attention and care to the patient. The questions have five possible answers: 0 = never, 1 = almost never, 2 = sometimes, 3 = quite often, and 4 = almost always. The total score ranges from 0 to 88 points, with 46 points or lower indicating no burden, moderate burden between 47 and 55 points, and intense burden with 56 points or more. The internal consistency of the Zarit Burden Interview has been found to be good, with Cronbach's α = 0.86.
The Low Back Pain Disability Scale (Oswestry) | 12 weeks
  Oswestry test is a self-administered questionnaire specific to low back pain that measures limitations in daily activities. It consists of 10 questions with 6 answer possible each. The internal consistency of the Oswestry test with Cronbach's α, = 0.82.

CONTACTS AND LOCATIONS:
Locations (1):
- Andalusian Public Health System, Granada, Spain

REFERENCES:
- [Derived] Prieto-Moreno R, Mora-Traverso M, Estevez-Lopez F, Molina-Garcia P, Ortiz-Pina M, Salazar-Gravan S, Cruz-Guisado V, Gago ML, Martin-Matillas M, Ariza-Vega P. Effects of the ActiveHip+ mHealth intervention on the recovery of older adults with hip fracture and their family caregivers: a multicentre open-label randomised controlled trial. EClinicalMedicine. 2024 Jun 7;73:102677. doi: 10.1016/j.eclinm.2024.102677. eCollection 2024 Jul. PMID 38911836
- See also: Related Info — http://52.208.219.206/